CLINICAL TRIAL: NCT04090099
Title: Ultrasound-GTrialuided Bilateral Erector Spina Block Versus Parasternal Block in Adult Cardiac Surgery: A Prospective, Randomized, Controlled Study.
Brief Title: Bilateral Erector Spina Block Versus Parasternal Block in Adult Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Yavuz Orak, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019/14-08
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Morphine Consumption; Pain, Postoperative
Keywords: Erector Spinae Block, Parasternal block, Cardiac surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (No Intervention): PCA (Patient controlled analgesia) and morphine consumption will be monitored in the postoperative period.
- Group ES (Erector Spina Plane) (Active Comparator): A high frequency (10-18 MHz) ultrasound linear probe covered with a sterile sheath will be placed 2 cm to the side of the T5 spinous process, first to the right or left. After demonstrating the T5 transverse process and the erector spinae muscle on top, the 22-gauge, 80 mm insulated Quincke-type needle will be inserted into the skin at an angle of about 30 degrees from the cranial to the caudal, using an in-plane technique. When the transverse process is touched, the needle is withdrawn and after a negative aspiration test with 0.5 mL of normal saline and after a hypo-echogenic display and hydrodissection, a local anesthetic solution will be applied to the fascia under the erector spinae muscle. A dose of 0.25% bupivacaine will be injected which is shown to spread both above and below the T5 level. The same process will be implemented on the other side.
  Interventions: Other: Erector spina plane block
- Group PS (Para Sternal Block) (Active Comparator): Before the wire is inserted into the sternum, the sternotomy and mediastinal tube regions will be infiltrated with a mixture of bupivacaine and saline.
  Interventions: Other: Erector spina plane block

INTERVENTIONS:
Other: Erector spina plane block — While the patient is in the sitting position, an area containing 2 cm lateral of the T5 spinous process will be cleaned with povidone iodine. A high frequency ultrasound linear probe covered with a sterile sheath will be placed 2 cm to the side of the T5 spinous process, first to the right or left. After demonstrating the T5 transverse process and the erector spinae muscle on top, the 22-gauge, 80 mm insulated Quincke-type needle will be inserted into the skin at an angle of about 30 degrees from the cranial to the caudal, using an in-plane technique. When the transverse process is touched, the needle is withdrawn and after a negative aspiration test with 0.5 mL of normal saline and after a hypo-echogenic display and hydrodissection, a local anesthetic solution will be applied to the fascia under the erector spinae muscle.
  Arms: Group ES (Erector Spina Plane); Group PS (Para Sternal Block)

SUMMARY:
Inadequate pain relief after cardiac surgery increases morbidity and results in a high incidence of persistent poststernotomy pain syndrome. The use of special opioid-based analgesia causes adverse effects such as nausea, vomiting, sedation, urinary retention, respiratory depression and delayed tracheal extubation. Regional anesthesia techniques such as pectoralis nerve block and serratus anterior block provide analgesia in the sternum and pain relief in the lateral / posterior chest Wall. Erector spinae (ESP) block, a new and simple myofascial block, provides wide multi-dermatomal sensory block. In the T5 spinous process, bilateral ESP block provides analgesia from T2 to T9 sensory level, resulting in both somatic and visceral analgesia by blocking both the dorsal and ventral of the spinal nerves, including the sympathetic chain. This block may provide adequate analgesia for median sternotomy because the main nerve supply to the sternal region is from T2 to T6. Median sternotomy incision and mediastinal tube regions are the major source of pain in patients undergoing cardiac surgery. The anterior and posterior branches of the intercostal nerves give nerves to the sternum. Parasternal local anesthetic infiltration around the sternum is effective in providing early postoperative analgesia and reducing opioid requirements and therefore has positive effects on healing. This simple and fast technique can be used even for anticoagulated patients.

DETAILED DESCRIPTION:
99 patients will be included in the study. Group C (Control, n = 31), Group ES (Erector Spina, n = 31), Group PS (Parasternal Intercostal Block n = 31) will be randomized. Randomization was achieved by randomly assigning patients to computer-generated random numbers. It will be explained that patients can receive both intravenous analgesia treatment and both blocks that are thought to be done. Patients will be told to express the degree of postoperative pain in the preoperative preparation room using a numerical scoring scale (NRS) between 0 and 10 (no pain at 0, no pain at 10). The vascular access will be opened in the pre-operative preparation room and 2 mg demizolam will be made. All preoperative cardiac drugs, except antiplatelet and anticoagulants, will be continued until the morning of surgery.

Demographic structures, cardiopulmonary bypass time, aortic cross clamp time, surgical time, ejection / fraction values will be recorded.

Weight and height of patients will be recorded (BMI). Preoperative, blood group and typing, full hemogram, liver function tests, renal function tests, chest radiography, electrocardiography, 2D transthoracic echocardiography and coronary angiography will be done as routine investigations.

Platelet count, bleeding time, clotting time, prothrombin time, activated partial thromboplastin time will be checked in all patients.

Constructional blocks:

1. ESP (Erector Spina Plane) Block Group
2. 2. Parasternal Block Group
3. Control Group The control group will not receive any Erector Spina block and Paravertebral Block. Only PCA (Patient Control Analgesia) and intravenous analgesic (Morphine) drug will be used.

The same surgical and anesthesia team will manage the patients. 6 channel ECG and non-invasive arterial pressure monitoring will be performed after the patients are admitted to the operation room. A peripheral intravenous line with a 16-gauge needle and a right radial artery with a 20-gauge needle will be performed. Blood will be taken for preoperative blood gas. Midazolam 0.01 (mg / kg), fentanyl (5-8 μg / kg) and rocuronium (0.6 mg / kg) will be used for induction of anesthesia. After anesthesia, central venous catheter and urinary catheter will be inserted. During general anesthesia Sevoflurane will be used in the air-oxygen mixture with a concentration of 50% oxygen. Normocapnic variation will be provided (PCO2 = 35-45). A rocuronium 0.6 mg / kg will be used every 30 minutes. All patients will undergo median sternotomy. Heparin 300-500 Units / kg to be administered. Activeted clotting time (ACT) will be kept> 400 throughout the procedure. Esophageal temperature will be monitored. The mean arterial pressure throughout the operation will be maintained above 60 mm Hg. Peroperative blood sample will be taken from the radial artery 3-5 minutes after the cross-clamp is removed. Heparin will be neutralized with protamine 1: 1.3. After the operation, patients will be transferred to the intensive care unit.

In the intensive care unit, patients will be extubated when the respiratory effort occurs, when the patient is awake, blood gas values are within normal range, body temperature is normal and hemodynamically stable. Morphine consumption by PCA and NRS scores will be monitored and recorded at 1, 3, 6, 12 and 24 hours after extübation. MAP (Mean arterial pressure), PH, PO2 (Blood gas) follow-ups will be recorded in the first blood gas, extubation and postoperative 1,2, 4,6,12, 24 hours.Paracetamol 1 g and Tramadol 1mg/kg intravenously will be administered to the patient if NRS> 3 when the patient is extubated.

If the patient's consciousness and hemodynamic status do not allow pain assessment, the patient will be excluded from the study. After the surgery, the investigator who evaluates NRS scores in the ICU will not know which group the patient is.

Oral feeding at postoperative hour, intensive care unit stay day, Side effects Nausea, Vomiting, Itching to be followed

ELIGIBILITY:
Inclusion Criteria:

* Male and / or female patients
* Aged 18-65 years
* Patients who will have coronary artery surgery under cardiopulmonary baypass (changing one, two and three vessels) with normal left ventricular function,
* Valve diseases with normal left ventricular function,
* ASD (Atrial Septal Defect) cases for atrial septal defect closure
* Patients with valve + CABG without left ventricular dysfunction will be included in the study.
* Ejection- Fraction> 50-55

Exclusion Criteria:

* Emergency and repeat heart surgery cases
* Advanced left coronary artery disease and left ventricular dysfunction
* Receiving preoperative inotropic support therapy,
* With mitral stenosis with atrial tombus,
* With low cardiac out put syndrome,
* Need intra-aortic balloon pump during surgery,
* Bleeding and coagulation disorder,
* Liver and kidney dysfunction,
* Patients with uncontrolled diabetes mellitus and coronary artery pulmonary disease,
* Opioid, analgesic and bupivacaine allergy,
* Patients with atrial fbrilation using anticoagulants
* Patients with cognitive dysfunction
* Patients who do not want to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Morphine consumption by PCA | Change from baseline 1 , 3, 6, 12 and 24 hours after extubation
  Morphine consumption used in case of pain

SECONDARY OUTCOMES:
Change Pain Scores | Time Frame: 1 hour,3 hours, 6 hours, 12 hours, 24 hours after the extubation
  NRS (Numeric Rating scale) Score. from 1 to 10 , 0: No pain, 10: 10 pain that can not be tolerated
Change Blood Gas | Change from Baseline at 60 minutes,2 hours, 4 hours, 6 hours, 12 hours, 24 hours after extübation ,
  PH, PO2
Blood Pressure | Change from Baseline at 60 minutes,2 hours, 4 hours, 6 hours, 12 hours, 24 hours after extübation ,
  mean arterial pressure mmHg

CONTACTS AND LOCATIONS:
Overall Officials: yavuz orak, md, Principal Investigator — Kahramanmaraş Sutcu Imam University Faculty of Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Kahramanmaras Sutcu Imam Univercity Faculty of edicine, Kahramanmaraş, Onikişubat
  - Kahramanmaras Sutcu Imam University Faculty of Medicine, Kahramanmaraş, Onikişubat

IPD SHARING:
Plan to Share IPD: No